CLINICAL TRIAL: NCT02593994
Title: Evaluation of Effectiveness and Safety of Resolute Onyx™ and Onyx Frontier™ in Routine Clinical Practice; A Multicenter, Prospective Observational Study
Brief Title: IRIS-Onyx Cohort in the IRIS-DES Registry
Acronym: IRIS-Onyx
Status: Active, not recruiting | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); Medtronic Korea Co., Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD, PhD, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2015-04
Record Dates: First submitted 2015-10-30; First posted 2015-11-02 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease; Arterial Occlusive Diseases; Cardiovascular Diseases; Percutaneous Transluminal Angioplasty
Keywords: Onyx; drug eluting stent; Routine Clinical Practice; Angioplasty, Transluminal, Percutaneous Coronary; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease; Arterial Occlusive Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Onyx Drug Eluting Stent
  Interventions: Device: Onyx Drug Eluting Stent group

INTERVENTIONS:
Device: Onyx Drug Eluting Stent group

SUMMARY:
The purpose of this study is to evaluate the relative effectiveness and safety of Onyx stent compared to other (drug eluting stents) DES.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and more
* Intervention with Onyx Drug Eluting Stent
* Agreed with written informed consent form

Exclusion Criteria:

* Intervention with Onyx drug eluting coronary stent and other drug eluting stent at the same time
* Life expectancy of 1year and under
* Cardiac shock

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Onyx Drug Eluting Stent
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Stent thrombosis | 1 year
  As per Academic Research Consortium (ARC) standard, definite or probable stent thrombosis

SECONDARY OUTCOMES:
All death | 5 year
Cardiac death | 5 year
Myocardial infarction | 5 year
Composite event of death or myocardial infarction | 5 year
Composite event of cardiac death or myocardial infarction | 5 year
Composite event rate | 5 year
  death, myocardial infarction, target vessel revascularization
Target Vessel revascularization | 5 year
Target Lesion revascularization | 5 year
Stent thrombosis | 5 year
Stroke | 5 year
Procedural success | 3 day
  defined as less than 30% residual stenosis at the completion of procedure without death or Q wave myocardial infarction or urgent revascularization participants will be followed for the duration of hospital stay, an expected average of 3days.

CONTACTS AND LOCATIONS:
Locations (31):
- South Korea (31):
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul, Republic of Korea
  - Asan Medical Center, Seoul, Songpa-gu
  - Hallym University Sacred Heart Hospital, Anyang
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Gangwon National Univ. Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - Inje University Ilsan Paik Hospital, Ilsan
  - Presbyterian Medical Center, Jeonju
  - Kwangju Christian Hospital, Kwangju
  - Dong-A Medical Center, Pusan
  - Inje University Pusan Paik Hospital, Pusan
  - Pusan National University Hospital, Pusan
  - Bundang CHA Hospital, Seongnam
  - Gangnam Severance Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea St. Paul's Hospital, Seoul
  - St.carollo Hospital, Suncheon
  - Ulsan University Hospital, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.